CLINICAL TRIAL: NCT04106583
Title: A Prospective, Multicenter Study Assessing the Embolization of Intracranial Aneurysms Using WAVE™ Extra Soft Coils, a Part of the Penumbra SMART COIL® System
Brief Title: Assessing the WAVE Extra Soft Coil in Intracranial Aneurysms and Comparing Imaging Modalities
Acronym: SURF
Status: Completed | Type: Observational
Sponsor: Penumbra Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CLP 13669
Record Dates: First submitted 2019-09-25; First posted 2019-09-27 (Actual); Results first posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Aneurysm, Brain
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Single Arm: Single Arm - Patients with intracranial aneurysms treated with WAVE, as part of the Penumbra SMART COIL System
  Interventions: Device: WAVE, as part of the SMART COIL System

INTERVENTIONS:
Device: WAVE, as part of the SMART COIL System — WAVE, as part of the SMART COIL System

SUMMARY:
The objective of this study is to demonstrate the safety and efficacy of the Penumbra SMART COIL® System, including the WAVE™ Extra Soft Coils (WAVE) as a fill and finish coil, in the treatment of intracranial aneurysms. Imaging will be analyzed by an independent core lab to assess aneurysm occlusion rates and perform a comparative analysis between imaging modalities.

ELIGIBILITY:
Inclusion Criteria:

* Patient age ≥ 18 years
* Patient having embolization of intracranial aneurysms
* WAVE Extra Soft Coil is final finishing coil
* Penumbra SMART COIL System accounts for at least 75% of total number of coils implanted
* Informed consent obtained per Institutional Review Board/Ethics Committee (IRB/EC) requirements

Exclusion Criteria:

* Life expectancy less than 1 year
* Patient previously enrolled in the SURF Study
* Known multiple intracranial aneurysms requiring treatment during index procedure
* Patient is unwilling or unable to comply with protocol follow up schedule and/or based on the Investigator's judgment the patient is not a good study candidate
* Participation in an interventional drug or device study that may confound the results of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with intracranial aneurysms treated with WAVE, as part of the Penumbra SMART COIL System
Sampling Method: Non-Probability Sample
Enrollment: 572 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2023-08-02 (Actual); Study Completion 2023-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clemens M Schirmer, MD, Principal Investigator — Geisinger Clinic
Locations (43):
- United States (34):
  - Southeast Health Medical Center, Dothan, Alabama
  - Banner UMC Tucson, Tucson, Arizona
  - Sharp Grossmont, La Mesa, California
  - Los Robles, Thousand Oaks, California
  - HRI - Swedish, Englewood, Colorado
  - St. Anthony's Hospital, Lakewood, Colorado
  - Yale New Haven, New Haven, Connecticut
  - University of Miami (Jackson Memorial), Miami, Florida
  - University of South Florida, Tampa, Florida
  - Morton Plant, Tampa, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Amita Health, Joliet, Illinois
  - Indiana University Health, Indianapolis, Indiana
  - Ochsner Medical Center, New Orleans, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Metro Health, Wyoming, Michigan
  - SSM Health Care, Bridgeton, Missouri
  - Northwell Health, Manhasset, New York
  - Mount Sinai Hospital, New York, New York
  - Westchester Medical Center, Valhalla, New York
  - Vidant Medical Center, Greenville, North Carolina
  - Mercy St. Vincent, Toledo, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Geisinger Medical Center, Danville, Pennsylvania
  - UPenn, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - MUSC, Charleston, South Carolina
  - Greenville Memorial Hospital, Greenville, South Carolina
  - University of Tennessee Medical Center, Knoxville, Knoxville, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - McAllen Medical Center, McAllen, Texas
  - Texas Stroke Institute - DFW, Plano, Texas
  - Riverside Regional Medical Center, Newport News, Virginia
- Canada (2):
  - Foothills Medical Center, Calgary
  - University Health Network, Toronto
- Germany (3):
  - Bremen-Mitte, Bremen
  - Klinikum Chemnitz gGmbH, Chemnitz
  - UKSH - Campus Lübeck, Lübeck
- Maggiore della Carità, Novara, Italy
- Spain (2):
  - Vall d'Hebron, Barcelona
  - Donostia, San Sebastián
- Universitätsspital Basel, Basel, Switzerland

REFERENCES:
- [Derived] Schirmer CM, Yoo AJ, Spiotta AM, Kaminsky I, Alshekhlee A, Starke RM, Nicholson A, Zaidat OO, Bohnstedt B, Psychogios MN, Viets R, Asif KS, Stapleton CJ, Mitha AP, Goren O; SURF Study Investigators. Intracranial aneurysm embolization using Penumbra fill and finish coils: 1-year results of a prospective, real-world, multicenter SURF study. J Neurointerv Surg. 2025 Sep 4:jnis-2025-023633. doi: 10.1136/jnis-2025-023633. Online ahead of print. PMID 40908130

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Arm
Started | 572
Completed | 494
Not Completed | 78

BASELINE CHARACTERISTICS:
Population: The analysis population consisted of the Intent-to-Treat (ITT) population that included all 572 enrolled patients. The primary analysis, including all effectiveness, safety, and subgroup reporting, were analyzed on this population.
Arm/Group | Single Arm
Number analyzed (Participants) | 572
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 356
  >=65 years | 216
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.5 (12.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 415
  Male | 157
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: 47 out of 572 participants were not analyzed due to data not collected in the EU.
  Participants
    number analyzed (Participants) | 525
    Hispanic or Latino | 79
    Not Hispanic or Latino | 389
    Unknown or Not Reported | 57
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 47 out of 572 participants were not analyzed due to data not being collected in the EU.
  27 out of the 525 analyzed participants were categorized as Race: "Other" - this number was added to 16 participants that were categorized under Race: "Unkown or Not Reported" in the Clinical Trial Report.
  Participants
    number analyzed (Participants) | 525
    American Indian or Alaska Native | 1
    Asian | 18
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 83
    White | 374
    More than one race | 6
    Unknown or Not Reported | 43
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] — Population: The analysis population (ITT) contains 558 evaluable participants.
  kg/m2
    number analyzed (Participants) | 558
    (all) | 28.6 (7.69)

OUTCOME MEASURES:

1. Primary Outcome: Efficacy: Adequate Occlusion
Description: Adequate occlusion defined as Raymond-Roy Class I and II at final follow-up
  Raymond-Roy Class grading ranges I to III higher values represent a worse outcome.
Time Frame: Through Study Completion, An Average of 1 Year
Population: The analysis population (ITT) contains 396 evaluable participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 396
Participants | 366

2. Primary Outcome: Safety: Serious Adverse Events (SAEs)
Description: The primary safety endpoints are SAEs within 24 hours post-procedure
Time Frame: Up to 24 Hours Post-Procedure
Population: The analysis population (ITT) contains 572 evaluable participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 572
Participants | 53

3. Primary Outcome: Safety: Device-Related SAE
Description: Device-related SAE up to 7 days or discharge
Time Frame: Through Discharge, up to 7 Days Post-Procedure
Population: The analysis population (ITT) contains 567 evaluable participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 567
Participants | 6

4. Secondary Outcome: Efficacy: Occlusion Rate
Description: Immediate post-procedure occlusion rates:
  Class 1 - Complete occlusion Class 2 - Residual neck Class 3 - Residual aneurysm
  The classification of angiographic results was adopted from Roy, Milot, and Raymond. Stroke 2001;32:1998-2004
Time Frame: Immediate Post-Procedure
Population: The analysis population (ITT) contains 570 evaluable participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 570
Participants
  Participants with Raymond-Roy Occlusion Class I | 361
  Participants with Raymond-Roy Occlusion Class II | 137
  Participants with Raymond-Roy Occlusion Class III | 72

5. Secondary Outcome: Efficacy: Retreatment Rate
Description: Retreatment rate at final follow-up
Time Frame: Through Study Completion, An Average of 1 Year
Population: The analysis population (ITT) contains 457 evaluable participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 457
Participants | 45

6. Secondary Outcome: Efficacy: Aneurysm Occlusion Raymond I
Description: Raymond-Roy Class grading ranges I to III higher values represent a worse outcome.
Time Frame: Immediate Post-Treatment
Population: The analysis population (ITT) contains 570 evaluable participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 570
Participants | 361

7. Secondary Outcome: Efficacy: Aneurysm Occlusion Raymond I
Description: Raymond-Roy Class grading ranges I to III higher values represent a worse outcome.
Time Frame: Through Study Completion, An Average of 1 Year
Population: The analysis population (ITT) contains 396 evaluable participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 396
Participants | 313

8. Secondary Outcome: Efficacy: Aneurysm Recanalization or Progressive Thrombosis
Description: Aneurysm recanalization or progressive thrombosis from post procedure to final follow-up
Time Frame: From Immediate Post Procedure Through Study Completion, An Average of 1 Year
Population: The analysis population (ITT) contains 395 evaluable participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 395
Participants
  Progressive Thrombosis | 110
  Stable Raymond-Roy Occlusion | 235
  Recanalization | 50

9. Secondary Outcome: Safety: Major Ipsilateral Stroke
Description: Occurrence of Major Ipsilateral Stroke
Time Frame: Through Study Completion, An Average of 1 Year
Population: The analysis population (ITT) contains 572 evaluable participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 572
Participants | 10

10. Secondary Outcome: Safety: Device-Related SAE
Description: Device related SAE at final follow-up
Time Frame: Through Study Completion, An Average of 1 Year
Population: The analysis population (ITT) contains 572 evaluable participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 572
Participants | 6

11. Secondary Outcome: Safety: Morbidity and Mortality
Description: All-cause morbidity and mortality at final follow-up
Time Frame: Through Study Completion, An Average of 1 Year
Population: The analysis population (ITT) contains 572 evaluable participants. Morbidity through Final Follow-Up was reported in 106 out of 572 participants, and One-Year Mortality was reported in 36 out of 572 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 572
Participants | 123

ADVERSE EVENTS:
Time Frame: Procedure, 7-day and/or Discharge, and final follow-up 1 year +/- 90 days
Description: In this study, only device-related or procedure-related adverse events and all serious adverse events (SAEs) were collected from procedure through discharge. After discharge, only neurological SAEs were collected. Additional information for Symptomatic Intracranial Hemorrhage and Ischemic Stroke will be collected on Event of Interest case report forms (CRF).
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 36/572
Serious Adverse Events (participants affected / at risk) | 140/572
Other Adverse Events (participants affected / at risk) | 20/572
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=572)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Cardiac arrest (Cardiac disorders) | 3 (3)
Cardiogenic shock (Cardiac disorders) | 1 (1)
Diabetes insipidus (Endocrine disorders) | 1 (1)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 4 (4)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 (1)
Cardiac death (General disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Death (General disorders) | 4 (4)
Infusion site haematoma (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Vascular stent occlusion (General disorders) | 1 (1)
Vascular stent thrombosis (General disorders) | 4 (4)
Anaphylactic reaction (Immune system disorders) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1)
Klebsiella sepsis (Infections and infestations) | 1 (1)
Meningitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 7 (7)
Pneumonia bacterial (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 5 (5)
Septic shock (Infections and infestations) | 2 (2)
Staphylococcal infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2)
Aneurysm perforation (Injury, poisoning and procedural complications) | 4 (4)
Burns second degree (Injury, poisoning and procedural complications) | 1 (1)
Device placement issue (Injury, poisoning and procedural complications) | 4 (4)
Mental status changes postoperative (Injury, poisoning and procedural complications) | 2 (2)
Subdural haematoma (Injury, poisoning and procedural complications) | 2 (2)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 2 (2)
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Weaning failure (Injury, poisoning and procedural complications) | 1 (1)
Angiogram cerebral abnormal (Investigations) | 1 (1)
Cerebral salt-wasting syndrome (Metabolism and nutrition disorders) | 2 (2)
Malnutrition (Metabolism and nutrition disorders) | 1 (1)
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Aphasia (Nervous system disorders) | 1 (1)
Brain compression (Nervous system disorders) | 2 (2)
Brain oedema (Nervous system disorders) | 3 (3)
Brain stem infarction (Nervous system disorders) | 1 (1)
Cerebellar microhaemorrhage (Nervous system disorders) | 1 (1)
Cerebral artery embolism (Nervous system disorders) | 2 (2)
Cerebral artery occlusion (Nervous system disorders) | 1 (1)
Cerebral artery thrombosis (Nervous system disorders) | 3 (3)
Cerebral infarction (Nervous system disorders) | 5 (5)
Cerebral venous sinus thrombosis (Nervous system disorders) | 1 (1)
Cerebrospinal fluid leakage (Nervous system disorders) | 1 (1)
Cytotoxic oedema (Nervous system disorders) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Embolic stroke (Nervous system disorders) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 4 (4)
Hemiparesis (Nervous system disorders) | 2 (2)
Hydrocephalus (Nervous system disorders) | 5 (5)
Intracranial aneurysm (Nervous system disorders) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 22 (24)
Loss of consciousness (Nervous system disorders) | 1 (1)
Migraine (Nervous system disorders) | 1 (1)
Neurological decompensation (Nervous system disorders) | 2 (2)
Posthaemorrhagic hydrocephalus (Nervous system disorders) | 4 (4)
Ruptured cerebral aneurysm (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 7 (8)
Stroke in evolution (Nervous system disorders) | 5 (5)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
VIth nerve paralysis (Nervous system disorders) | 1 (1)
Device dislocation (Product Issues) | 1 (1)
Mental status changes (Psychiatric disorders) | 2 (4)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Aneurysm repair (Surgical and medical procedures) | 1 (1)
Cerebral oedema management (Surgical and medical procedures) | 1 (1)
Reduction of increased intracranial pressure (Surgical and medical procedures) | 1 (1)
Surgery (Surgical and medical procedures) | 1 (1)
Ventriculo-peritoneal shunt (Surgical and medical procedures) | 1 (1)
Aneurysm ruptured (Vascular disorders) | 1 (1)
Aortic dissection (Vascular disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 3 (3)
Embolism (Vascular disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Peripheral artery stenosis (Vascular disorders) | 1 (1)
Thrombosis (Vascular disorders) | 4 (4)
Vascular dissection (Vascular disorders) | 1 (1)
Vasoconstriction (Vascular disorders) | 1 (1)
Vasospasm (Vascular disorders) | 42 (46)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=572)
Pain (General disorders) | 1 (1)
Vascular stent thrombosis (General disorders) | 1 (1)
Aneurysm perforation (Injury, poisoning and procedural complications) | 3 (3)
Procedural vomiting (Injury, poisoning and procedural complications) | 1 (1)
Vascular access site haematoma (Injury, poisoning and procedural complications) | 1 (1)
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Vascular access site pain (Injury, poisoning and procedural complications) | 1 (1)
Cerebral artery embolism (Nervous system disorders) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1)
Cerebral reperfusion injury (Nervous system disorders) | 1 (1)
Embolic cerebral infarction (Nervous system disorders) | 2 (2)
Embolic stroke (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Peripheral artery occlusion (Vascular disorders) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)
Vasospasm (Vascular disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-01): https://cdn.clinicaltrials.gov/large-docs/83/NCT04106583/Prot_SAP_000.pdf